CLINICAL TRIAL: NCT05968807
Title: "The Isolation I Feel is Profound": The iParent2Parent Online Peer Support Program for Parents of Pediatric Solid Organ Transplantation Recipients
Brief Title: iParent2Parent Program for Parents of Pediatric Solid Organ Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Samantha Anthony, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000080779
Record Dates: First submitted 2023-06-29; First posted 2023-08-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Solid Organ Transplant
Keywords: Peer Support Mentorship; Parent Support Mentorship; Pediatrics; Transplant

STUDY DESIGN:
Intervention Model Description: Waitlist randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iParent2Parent Program (Experimental)
  Interventions: Behavioral: iParent2Parent Program
- Standard of Care Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: iParent2Parent Program — iParent2Parent is an online peer support mentorship program that is based on the iPeer2Peer online peer support mentorship program, which has been established in multiple chronic disease populations as a self-management intervention, including in chronic pain and juvenile idiopathic arthritis populations. The iParent2Parent program connect parents one-to-one with other parents of pediatric solid organ transplant (SOT) recipients who are trained to offer vital peer support and mentorship.
  Arms: iParent2Parent Program

SUMMARY:
The iParent2Parent (iP2P) program is a new, innovative virtual mentorship program that will connect parents one-to-one with other parents of pediatric solid organ transplant (SOT) recipients who are trained to offer vital peer support and mentorship. Parents of children who received a SOT at The Hospital for Sick Children will be invited to participate as mentors and mentees (randomized into the iP2P or control group). The iP2P program can decrease feelings of isolation, improve mental health and have a long-term positive impact on patient health. This research will increase our understanding of one-to-one peer support and leverage eHealth technologies to improve the access to and acceptability of parent peer support interventions.

ELIGIBILITY:
Mentee Inclusion Criteria:

* Parent of a patient under 18 years of age who received a solid organ transplant and is at least two months post-transplant,
* Access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software, and
* English-speaking.

Mentor Inclusion Criteria:

* Parent of a patient under 21 years of age who received a solid organ transplant and is at least one year post-transplant,
* Nominated by their child's healthcare team as a good candidate to act in the mentor role (e.g., good communication skills, positive adaptation and adjustment post-transplant, strong support network),
* Access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software, and
* English-speaking.

Exclusion Criteria:

* Non-English speaking.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates and withdrawal rates | Baseline to study completion, an average of 1 year
  How many participants were recruited and have withdrawn from the program on average over time.
Adherence with the iParent2Parent program | Baseline to study completion, an average of 1 year
  When the participant completes 10 audio or video calls over 12 weeks and 100% when all online outcome measures completed.
Acceptability (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Whether the innovation is agreeable, palatable or satisfactory.
  Measured via semi-structured interview or focus group.
Acceptability (Mentors) | Baseline to program completion, an average of one year
  Whether the innovation is agreeable, palatable or satisfactory.
  Measured via semi-structured interview or focus group.
Level of engagement with the iParent2Parent program (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Measured via semi-structured interview or focus group.
Level of engagement with the iParent2Parent program (Mentors) | Baseline to program completion, an average of one year
  Measured via semi-structured interview or focus group.
Barriers and enablers of the iParent2Parent program (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Measured via semi-structured interview or focus group.
Barriers and enablers of the iParent2Parent program (Mentors) | Baseline to program completion, an average of one year
  Measured via semi-structured interview or focus group.

SECONDARY OUTCOMES:
Parenting stress (Mentees and Mentors) | Baseline to program completion, an average of one year
  Parental Stress Scale; 18-item questionnaire. Each question is scored on a scale from 1 to 5, with scores ranging from 18 to 90. An overall higher score means a worse outcome.
Psychological distress (Mentees and Mentors) | Baseline to program completion, an average of one year
  General Anxiety Disorder-7; 7-item questionnaire. Each question is scored on a scale from 0 to 3, with scores ranging from 0 to 21. An overall higher score means a worse outcome.
Psychological distress (Mentees and Mentors) | Baseline to program completion, an average of one year
  Patient Health Questionnaire Depression Scale; 8-item questionnaire. Each question is scored on a scale from 0 to 3, with scores ranging from 0 to 24. An overall higher score means a worse outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Social Isolation; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a worse outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Informational Support; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a better outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Emotional Support; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a better outcome.
Coping (Mentees and Mentors) | Baseline to program completion, an average of one year
  Coping Health Inventory for Parents; 16-item questionnaire. Each question about coping behaviour is scored on a scale from 0 to 3, with a possible response of "Did not use" the coping behaviour. Scores range from 0 to 48. An overall higher score means a better outcome.
Family Functioning (Mentees and Mentors) | Baseline to program completion, an average of one year
  Pediatric Quality of Life Inventory™ 2.0 Family Impact Module; 36-item questionnaire with 8 different sections: Physical Functioning, Emotional Functioning, Social Functioning, Cognitive Functioning, Communication, Worry, Daily Activities, and Family Relationships. Each question is scored on a scale from 0 to 4. Items are reverse-scored and linearly transformed to a 0-100 scale. An overall higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J. Anthony, PhD, MSW, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No